CLINICAL TRIAL: NCT00418392
Title: Intrapleural Minocycline After Simple Aspiration for the Prevention of Primary Spontaneous Pneumothorax: A Randomized Trial
Brief Title: Intrapleural Minocycline After Simple Aspiration for the Prevention of Primary Spontaneous Pneumothorax
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 950510; DOH95-TD-I-111-012
Record Dates: First submitted 2006-12-31; First posted 2007-01-04 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-11

CONDITIONS: Pneumothorax
Keywords: pneumothorax, aspiration, minocycline, pleurodesis
MeSH Terms: conditions — Pneumothorax; cyclopia sequence

ARMS (2):
- Minocycline group (Experimental): After successful simple aspiration, minocycline pleurodesis will be performed.
  Interventions: Procedure: Simple aspiration with minocycline pleurodesis
- Control group (Placebo Comparator): After successful simple aspiration, nothing will be performed.
  Interventions: Procedure: simple aspiration

INTERVENTIONS:
Procedure: Simple aspiration with minocycline pleurodesis — Intrapleural instillation of 300mg minocycline within 5 min after simple aspiration
  Arms: Minocycline group
Procedure: simple aspiration — Simple aspiration for primary spontaneous pneumothorax by pigtail catheter
  Arms: Control group

SUMMARY:
The estimated recurrence rate of primary spontaneous pneumothorax is 23-50% after the first episode, and the optimal treatment remains unknown. In the recently published British Thoracic Society (BTS) guidelines, simple aspiration is recommended as first line treatment for all primary pneumothoraces requiring intervention. However, the 1 year recurrence rate of this procedure was as high as 25-30%, making it inappropriate as a standard of care.

Intrapleural instillation of a chemical irritant (chemical pleurodesis) is an effective way to shorten the duration of air leaks and reduce the rates of recurrent spontaneous pneumothorax in surgical and non-surgical patients. Many chemical irritants (tetracycline, talc, and minocycline) have been used to decrease the rate of recurrence in spontaneous pneumothorax. Tetracycline, which was the most commonly used irritant, is no longer available. Talc insufflation of the pleural cavity is safe and effective for primary spontaneous pneumothorax. However, it should be applied either with surgical or medical thoracoscopy. Minocycline, a derivative of tetracycline, is as effective as tetracycline in inducing pleural fibrosis in rabbits. In the previous studies, we have shown that additional minocycline pleurodesis is a safe and convenient procedure to decrease the rates of ipsilateral recurrence after thoracoscopic treatment of primary spontaneous pneumothorax. In the present study, additional minocycline pleurodesis will be randomly administered in patients with first episode of primary spontaneous pneumothorax after simple aspiration to test if it can reduce the rate of recurrence.

DETAILED DESCRIPTION:
Background:

Primary spontaneous pneumothorax most commonly occurs in young, tall, lean males (1, 2). The estimated recurrence rate is 23-50% after the first episode (3). Optimal treatment of patients presenting with a first episode of primary spontaneous pneumothorax remains unknown. In the recently published British Thoracic Society (BTS) guidelines (4), simple aspiration is recommended as first line treatment for all primary pneumothoraces requiring intervention. However, the 1 year recurrence rate of this procedure was as high as 26-30% (5), making it inappropriate as a standard of care.

Intrapleural instillation of a chemical irritant (chemical pleurodesis) is an effective way to shorten the duration of air leaks and reduce the rates of recurrent spontaneous pneumothorax in surgical and non-surgical patients (6, 7). Light et al. has shown that intrapleural tetracycline is effective in reducing the rate of ipsilateral recurrence for patients with spontaneous pneumothorax (7). However, the recently published guidelines recommended that chemical pleurodesis should only be attempted if the patient is either unwilling or unable to undergo surgery because the rates of recurrence of pneumothoraces after surgical intervention either by thoracotomy or VATS, with or without surgical pleurodesis, is far less than after chemical pleurodesis (4, 8). As a result, chemical pleurodesis has rarely been used in primary spontaneous pneumothorax, and the effect of additional chemical pleurodesis after simple aspiration in preventing recurrence of pneumothoraces has never been evaluated.

Tetracycline, which was the most commonly used irritant, is no longer available. Minocycline, a derivative of tetracycline, is as effective as tetracycline in inducing pleural fibrosis in rabbits (9). In the previous studies, we have shown that additional minocycline pleurodesis is a safe and convenient procedure that associates with lower rates of prolonged air leaks and ipsilateral recurrence after thoracoscopic treatment of primary spontaneous pneumothorax (10, 11).

In the present study, additional minocycline pleurodesis will be randomly administered in patients with first episode of primary spontaneous pneumothorax after simple aspiration to test if it can reduce the rate of recurrence. This study will comply with the protocol, GCP and applicable requirement of the Institutional Review Boards (IRB) of the NTUH and Far Eastern Memorial Hospital.

Patients and Methods:

Study design This study is a prospective, randomized, controlled trial to evaluate if additional minocycline pleurodesis after simple aspiration will be effective in preventing recurrence of primary spontaneous pneumothorax.

Primary Objective The primary end point is to compare the rates of ipsilateral recurrence between the minocycline and observation groups after simple aspiration of the pneumothorax.

Secondary Objectives

1. Safety profile of minocycline pleurodesis
2. Early results, including immediate success rates, one-week success rates, complication rates, rates of hospitalization, duration of hospitalization, and the degrees of chest pain.
3. Long-term effects of minocycline pleurodesis, including degrees of residual chest pain and pulmonary function test.

Eligibility criteria

Patients must meet ALL of the inclusion criteria for the entry of this study:

1. Male or female.
2. Age between 15 and 40 years old.
3. First episode of spontaneous pneumothorax.
4. Symptomatic (dyspnea or chest pain) or the rim of air is > 2cm on CXR requiring simple aspiration
5. Complete or nearly complete and persistent lung expansion immediately following manual aspiration
6. Organ Function Requirements:

   1. Adequate hematological function (Hb > 10 g/dl, ANC > 1.5 x 109/L, platelets > 100 x 109/L)
   2. Normal renal and hepatic functions: serum creatinine < 1 x ULN, SGPT and SGOT< 2.5 x ULN, alkaline phosphatase < 5 x ULN
7. Written inform consent

The exclusion criteria are:

1. With underlying pulmonary disease (asthma, chronic obstructive pulmonary disease, bronchiectasis, etc)
2. With hemothorax or tension pneumothorax requiring chest tube insertion or operation
3. A history of previous pneumothorax
4. A history of previous ipsilateral thoracic operation
5. Allergy to tetracycline or minocycline
6. Pregnant or lactating patients.
7. Other serious concomitant illness or medical conditions:

   1. Congestive heart failure or unstable angina pectoris.
   2. History of myocardial infarction within 1 year prior to the study entry.
   3. Uncontrolled hypertension or arrhythmia.
   4. History of significant neurologic or psychiatric disorders, including dementia or seizure.
   5. Active infection requiring i.v. antibiotics. Subjects who are unwilling to undergo randomization, treatment, or follow-up procedures will be removed from the study. Subjects can also withdraw from the trial at any time point by their will.

Randomization:

Patients will be randomized at each center with separate random number lists into one of the two treatment groups using a computer-generated table numerically corresponding with the treatment group. The trial treatment randomization codes will be maintained until the end of the study and will be broken by investigators who were blind to the randomization procedure.

Manual aspiration Manual aspiration will be performed as follows: patients were seated in semi-supine position. After skin disinfection and field preparation, a small-caliber pig-tail catheter (6-10 French) will be introduced after local anesthesia with 2% lidocaine in the second intercostal space, at the midclavicular line. After the catheter enters the pleural space, the catheter will be fixed to the skin using sterile adhesive tape and connected via a three-way valve to a 50-ml syringe. Air will be manually aspirated, until a resistance was felt and air was no longer aspirated. Thereafter, a chest X-ray will be performed with the catheter in place.

Minocycline pleurodesis In the minocycline group, 30 mL of 1% lidocaine hydrochloride (300mg) followed by a solution of 30 mL of normal saline containing 300 mg of minocycline (Mirosin®, Taiwan Panbiotic Laboratories, Kaohsiung, Taiwan) will be instilled into the pleural cavity through the pig-tail catheter or chest tube. In the observation group, nothing will be administered. Administration of other chemical pleurodesis agents is prohibited during the study period. Intramuscular meperidine hydrochloride (Demerol®, 50mg/ampule) will be administered every 4 to 6 hours according to the patient's request if the pain became intolerable, could not be relieved by oral analgesics, and visual analogue scale was greater than 7. Chest radiography will be performed immediate postoperatively or the next morning. VAS will be evaluated immediately 6 hours later after minocycline administration.

Study Endpoints:

The primary end point will be rate of ipsilateral recurrence after the procedure. Secondary end points include safety, early results, and long-term effects of minocycline pleurodesis.

Immediate success rates: defined as complete or nearly complete and persistent lung expansion immediately following manual aspiration. Immediate success for chest tube drainage is defined as complete lung expansion, absence of air leakage, and chest drain removal within 24 hours after catheter placement.

One weeks success rates are defined as complete and persistent lung expansion at one weeks after the first attempt of aspiration or tube insertion.

One-year success: absence of recurrent pneumothorax during a 1-year follow-up period. .

Safety assessments:

Safety assessments will consist of monitoring and recording all toxicity, adverse events, safety laboratory examination, vital signs, physical examination. The adverse events which are not reported will be graded as mild, moderate, severe, and life-threatening. Adverse event will be tabulated and the incidence rates will be calculated.

Sample size estimation:

A sample size of 300 patients (150 in each group) will be needed to reach clinical significance (at the .05 level with a power of 0.9) if minocycline reduced the recurrence rate from 30% to 15% and the drop out rate is 10%. A planned interim analysis will be conducted after enrollment of 150 patients with at least 12 months of follow-up. Statistical analysis will be performed on an intent-to-treat basis rather than in an actual treatment basis.

Follow-up After discharge from the hospital, patients will be followed at the outpatient clinics at 1 week, 1 month, 3 months, and 6 months where chest radiography will be performed. Follow-ups will then be conducted every 6 months by a registered nurse who is blinded to the group allocation by telephone conversation, according to a standard questionnaire that included when the patient returns to work or school, whether a recurrence occurred, when it happened, and how it is treated. Residual postoperative chest pain will be evaluated on a pain score from 0 to 5, where 0 is pain free; 1 is occasional discomfort; 2 is occasional use of analgesics; 3 is using nonopiate analgesics; 4 is regular pain using opiates; 5 is severe and intractable pain. All patients will be followed for at least 12 months. Patients can come back to the clinic or visit emergency department whenever they have chest pain, dyspnea, or any signs related to the recurrence of pneumothorax.

Pulmonary function analysis Pulmonary function tests will be performed for patients able to attend a hospital outpatient appointment at least 6 months after surgery. Forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1.0) will be measured using a spirometer of Microspiro HI-298 (Chest Corporation, Tokyo, Japan) with the patients seated. A minimum of three acceptable forced expiratory maneuvers will be performed and the best one will be selected for analysis.

Data collection and statistical analysis The clinical data, duration of chest drainage, length of hospital stay, complications, requested doses of meperidine, and data of VAS will be collected. Continuous variables such as age or weight will be expressed as the mean + standard deviation and analyzed by the two sample t-test. Categorical variables such as gender or smoking status will be presented by frequency (%) and analyzed by the Fisher's exact test. Intensity of postoperative pain measured by VAS (from 0 to 10) were summarized by mean (95 percent confidence interval) and compared by Wilcoxon rank-sum test. Scores of residual chest pain will be analyzed by the Wilcoxon rank-sum test. Freedom from recurrence will be analyzed by the Kaplan-Meier method, and comparisons will be made by the log-rank test.

Reference:

1. Gobbel WG Jr, Rhea WG, Nelson IA, Daniel RA Jr. Spontaneous pneumothorax. J Thorac Cardiovasc Surg 1963;46:331-345.
2. Lichter J, Gwynne JF. Spontaneous pneumothorax in young subjects. Thorax 1971;25:409-417.
3. Light RW. Management of spontaneous pneumothorax. Am Rev Respir Dis 1993;148:245-258.
4. Henry M, Arnold T, Harvey J; Pleural Diseases Group, Standards of Care Committee, British Thoracic Society. BTS guidelines for the management of spontaneous pneumothorax. Thorax 2003;58(Supple 2):39-52.
5. Noppen M, AJRCCM, 2003
6. Hatta T, Tsubota N, Yoshimura M, Yanagawa M. Intrapleural minocycline for postoperative air leakage and control of malignant pleural effusion. Kyobu Geka 1990;43:283-286.
7. Light RW, O'Hara VS, Moritz TE, McElhinney AJ, Butz R, Haakenson CM, Read RC, Sassoon CS, Eastridge CE, Berger R, et al. Intrapleural tetracycline for the prevention of recurrent spontaneous pneumothorax. JAMA 1990;264:2224-2230.
8. Baumann MH, Strange C, Heffner JE, Light R, Kirby TJ, Klein J, Luketich JD, Panacek EA, Sahn SA; AACP Pneumothorax Consensus Group. Management of spontaneous pneumothorax: an American College of Chest Physicians Delphi consensus statement. Chest 2001;119:590-602.
9. Light RW, Wang NS, Sassoon CSH, Gruer SE, Vargas FS. Comparison of the effectiveness of tetracycline and minocycline as pleural sclerosing agents in rabbits. Chest 1994;106:577-582.
10. Chen JS, Hsu HH, Kuo SW, Tsai PR, Chen RJ, Lee JM, Lee YC: Effects of additional minocycline pleurodesis after thoracoscopic procedures for primary spontaneous pneumothorax. Chest 2004;125:50-55.
11. Chen JS, Hsu HH, Chen RJ, Kuo SW, Huang PM, Tsai PR , Lee JM, Lee YC: Additional minocycline pleurodesis after thoracoscopic surgery for primary spontaneous pneumothorax. Am J Respir Crit Care Med 2006;173: 548-554.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Age between 15 and 40 years old.
3. First episode of spontaneous pneumothorax.
4. Symptomatic (dyspnea or chest pain) or the rim of air is > 2cm on CXR requiring simple aspiration
5. Complete or nearly complete and persistent lung expansion immediately following manual aspiration
6. Organ Function Requirements:

   * Adequate hematological function (Hb > 10 g/dl, ANC > 1.5 x 109/L, platelets > 100 x 109/L)
   * Normal renal and hepatic functions: serum creatinine < 1 x ULN, SGPT and SGOT< 2.5 x ULN, alkaline phosphatase < 5 x ULN
7. Written inform consent

Exclusion Criteria:

1. With underlying pulmonary disease (asthma, chronic obstructive pulmonary disease, bronchiectasis, etc)
2. With hemothorax or tension pneumothorax requiring chest tube insertion or operation
3. A history of previous pneumothorax
4. A history of previous ipsilateral thoracic operation
5. Allergy to tetracycline or minocycline
6. Pregnant or lactating patients.
7. Other serious concomitant illness or medical conditions:

   * Congestive heart failure or unstable angina pectoris.
   * History of myocardial infarction within 1 year prior to the study entry.
   * Uncontrolled hypertension or arrhythmia.
   * History of significant neurologic or psychiatric disorders, including dementia or seizure.
   * Active infection requiring i.v. antibiotics.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-11; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
to compare the rates of ipsilateral recurrence between the minocycline and observation groups after simple aspiration of the pneumothorax. | 12 months after treatment

SECONDARY OUTCOMES:
Safety profile of minocycline pleurodesis | 12 months after treatment
Early results, including immediate success rates, one-week success rates, complication rates, rates of hospitalization, duration of hospitalization, and the degrees of chest pain. | 7 days after treatment
Long-term effects of minocycline pleurodesis, including degrees of residual chest pain and pulmonary function test | 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Chie Lee, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Chen JS, Hsu HH, Chen RJ, Kuo SW, Huang PM, Tsai PR, Lee JM, Lee YC. Additional minocycline pleurodesis after thoracoscopic surgery for primary spontaneous pneumothorax. Am J Respir Crit Care Med. 2006 Mar 1;173(5):548-54. doi: 10.1164/rccm.200509-1414OC. Epub 2005 Dec 15. PMID 16357330
- [Background] Chen JS, Hsu HH, Kuo SW, Tsai PR, Chen RJ, Lee JM, Lee YC. Effects of additional minocycline pleurodesis after thoracoscopic procedures for primary spontaneous pneumothorax. Chest. 2004 Jan;125(1):50-5. doi: 10.1378/chest.125.1.50. PMID 14718420
- [Background] Light RW, O'Hara VS, Moritz TE, McElhinney AJ, Butz R, Haakenson CM, Read RC, Sassoon CS, Eastridge CE, Berger R, et al. Intrapleural tetracycline for the prevention of recurrent spontaneous pneumothorax. Results of a Department of Veterans Affairs cooperative study. JAMA. 1990 Nov 7;264(17):2224-30. PMID 2214100
- [Background] Henry M, Arnold T, Harvey J; Pleural Diseases Group, Standards of Care Committee, British Thoracic Society. BTS guidelines for the management of spontaneous pneumothorax. Thorax. 2003 May;58 Suppl 2(Suppl 2):ii39-52. doi: 10.1136/thorax.58.suppl_2.ii39. No abstract available. PMID 12728149
- [Derived] Chen JS, Chan WK, Tsai KT, Hsu HH, Lin CY, Yuan A, Chen WJ, Lai HS, Yang PC. Simple aspiration and drainage and intrapleural minocycline pleurodesis versus simple aspiration and drainage for the initial treatment of primary spontaneous pneumothorax: an open-label, parallel-group, prospective, randomised, controlled trial. Lancet. 2013 Apr 13;381(9874):1277-82. doi: 10.1016/S0140-6736(12)62170-9. Epub 2013 Mar 12. PMID 23489754